CLINICAL TRIAL: NCT05673291
Title: Evaluation of the Relationship Between Posture and Musculoskeletal Pain in Dentists
Brief Title: Posture and Musculoskeletal Pain in Dentists
Acronym: Pain
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, PhD,Akdeniz University, Physiotherapy Department, Akdeniz University
Other Study IDs: Akdeniz University Dentistry
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-01

CONDITIONS: Musculoskeletal Pain; Postural Kyphosis; Spinal Instability
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active working group: For the study group, dentists who have completed at least 1 year in the profession, actively working in their professional life, and 4th and 5th-year of intern dentistry students
  Interventions: Other: No intervention
- Control group: In the study, 3rd-grade dentistry students who have not yet started the clinical education process will be selected as the control group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Volunteers who will be included in the research will be informed about the research and an informed consent form will be signed. Questionnaire evaluating sociodemographic characteristics and working positions; The Extended Nordic Musculoskeletal Questionnaire (7) and measurements made with the Spinal Mouse device for posture analysis will be applied when individuals feel comfortable. Questionnaires and device and posture analysis will be carried out after the purpose of the research is explained to the individuals and their consent is obtained. The data will be analyzed in the SSPS program. Number, percentage, standard deviation and mean from descriptive statistics will be used in the evaluation of the data. The relationship between posture and musculoskeletal pain will be evaluated by correlation analysis. The confidence interval of the research will be 95% and the significance level will be considered as p<0.05.

SUMMARY:
Objectives: Musculoskeletal problems have been a concern in dentists for years. The aim of this study is to evaluate the relationship between posture and musculoskeletal pain in dentists.

DETAILED DESCRIPTION:
Working in an extremely challenging posture, performing movements that require force, and sitting or standing for a long time during dental practices are effective in the formation of musculoskeletal pain. Musculoskeletal pain; is caused by disorders affecting anatomical structures that provide structural support to our body, such as muscles, tendons, ligaments, cartilage, bones, and joints. Literature information shows that an average of 64% to 93% of dentists complain of musculoskeletal pain throughout their professional life.

Dentists often exhibit a negative posture characterized by neck flexion and shoulder abduction in order to provide a better field of view when treating their patients. Flattening of the cervical lordosis due to forward bending of the head and neck; Over time, it causes fatigue in the muscles in the neck and shoulder region, decrease in blood flow, pain, and ultimately protective muscle contractions. These irregularities in the muscles due to repetitive cumulative traumas can increase the force on the spinal discs of the neck and cause inevitable musculoskeletal diseases in the future. Similarly, a decrease in lumbar lordosis, right lateral flexion of the lumbar vertebrae, and leftward tilt of the thoracic vertebrae are characteristic positions during patient treatment in physicians who constantly sit and work, and studies have shown that there is a positive and significant correlation between this position and low back pain.

According to the definition of the Posture Committee of the American Academy of Orthopedic Surgeons, posture is the balanced and proper arrangement of skeletal elements in order to protect the body from deformations and prevent injury. Physiologically and biomechanically good posture is a posture that provides maximum efficiency in the body with minimum effort. It is important for a good posture that the four basic curvatures of the human spine, known as cervical and lumbar lordosis, thoracic and sacral kyphosis, are in harmony. Improper postural posture; accelerates the wear and tear in the vertebrae, discs, muscles, and ligaments, which causes pain. Therefore, the evaluation of posture is important in dentists.

Even in the best working position, dentists must have more than 50 muscles active in order to keep their body positions stable against gravity. Physicians generally lose their postural awareness during treatment shortly after starting treatment. During the treatment, they work in an inappropriate posture for a long time, neglecting their own health, mostly considering the treatment applications and the comfort of the patients. It is very important for physicians to be aware of the factors that cause musculoskeletal system problems and to learn to work in the right posture in order to maintain their health and practice their profession for a long time.

Posture evaluation of individuals is evaluated based on some reference points in the body. In this way, the relationship of body parts with each other and with gravity is compared with normal anatomical features, and deviations and differences are determined. The gold standard method in standard posture analysis is radiographic analysis. However, the use of radiography is undesirable due to the radiation it contains. The Spinal Mouse, which is an important tool in the measurement of posture correctness, is a device with mouse-shaped wheels that detects the angles and position of the spine and transfers them to the computer environment without the need for radiography and is a safe and non-invasive tool. It detects the curvature of the spine, its anatomical structure, and movements in the sagittal and frontal planes. It is an easy-to-use, fast and practical measuring device. Compared to radiography, it is important that it does not contain radiation and is non-invasive. The reliability and validity studies of the device have been carried out, and it provides quantitative data in order to obtain quick information about the posture. The raw data of the wireless and handheld mouse is transferred to the computer via Bluetooth and the data is evaluated in the computer environment. In this study, it is planned to obtain quantitative data about the postures of dentists by using the spinal mouse. In the literature review, only one study reported that there was a positive correlation between spinal mouse data and musculoskeletal pain in the evaluation of 1st, 3rd, and 5th-grade students using a spinal mouse. However, there is no study that evaluates the relationship between working hours, working positions, posture, and musculoskeletal pain in dentists working in different departments and compares them with the data of dentistry students who have just started their profession.

In light of all this information, the aim of this study is to evaluate the relationship between posture and musculoskeletal pain in dentists.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteered to participate in the study
* Dentists who have completed at least 1 year in the profession for the study group and are actively working in their professional life
* 4th and 5th year intern students
* 3rd-year students who do not do clinical training (Control group)

Exclusion Criteria:

* Congenital musculoskeletal disorder
* Having undergone musculoskeletal surgery
* Having a rheumatic or neurological disease
* Being pregnant

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dentistry 3-4-5th year students and dentists
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Sociodemographic data | 1-3 monts
  Questionnaire including sociodemographic characteristic
Extended Nordic Musculoskeletal Questionnaire,Spinal Mouse. | 1-3 months
  Assessing working posistions,Evaluation of posture with the Spinal Mouse device

SECONDARY OUTCOMES:
Goniometer assessment | 1-3 motnhs
  Evaluation of neck joint movements with goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Daltaban, PhD, Study Director — Akdeniz University Dentistry
Locations (1):
- Akdeniz Universitesi, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayes M, Cockrell D, Smith DR. A systematic review of musculoskeletal disorders among dental professionals. Int J Dent Hyg. 2009 Aug;7(3):159-65. doi: 10.1111/j.1601-5037.2009.00395.x. PMID 19659711
- [Background] Ng A, Hayes MJ, Polster A. Musculoskeletal Disorders and Working Posture among Dental and Oral Health Students. Healthcare (Basel). 2016 Jan 23;4(1):13. doi: 10.3390/healthcare4010013. PMID 27417601
- [Background] Mannion AF, Knecht K, Balaban G, Dvorak J, Grob D. A new skin-surface device for measuring the curvature and global and segmental ranges of motion of the spine: reliability of measurements and comparison with data reviewed from the literature. Eur Spine J. 2004 Mar;13(2):122-36. doi: 10.1007/s00586-003-0618-8. Epub 2003 Dec 6. PMID 14661104
- [Background] Csuhai EA, Nagy AC, Varadi Z, Veres-Balajti I. Functional Analysis of the Spine with the Idiag SpinalMouse System among Sedentary Workers Affected by Non-Specific Low Back Pain. Int J Environ Res Public Health. 2020 Dec 11;17(24):9259. doi: 10.3390/ijerph17249259. PMID 33322248
- [Background] Ripani M, Di Cesare A, Giombini A, Agnello L, Fagnani F, Pigozzi F. Spinal curvature: comparison of frontal measurements with the Spinal Mouse and radiographic assessment. J Sports Med Phys Fitness. 2008 Dec;48(4):488-94. PMID 18997653
- [Background] Kapitan M, Pilbauerova N, Vavrickova L, Sustova Z, Machac S. Prevalence of Musculoskeletal Disorders Symptoms Among Czech Dental Students. Part 2: The Predictive Value of Digital Assessment. Acta Medica (Hradec Kralove). 2019;62(1):6-11. doi: 10.14712/18059694.2019.39. PMID 30931890
- [Background] Dawson AP, Steele EJ, Hodges PW, Stewart S. Development and test-retest reliability of an extended version of the Nordic Musculoskeletal Questionnaire (NMQ-E): a screening instrument for musculoskeletal pain. J Pain. 2009 May;10(5):517-26. doi: 10.1016/j.jpain.2008.11.008. Epub 2009 Apr 2. PMID 19345154
- [Background] Kellis E, Adamou G, Tzilios G, Emmanouilidou M. Reliability of spinal range of motion in healthy boys using a skin-surface device. J Manipulative Physiol Ther. 2008 Oct;31(8):570-6. doi: 10.1016/j.jmpt.2008.09.001. PMID 18984239
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343